CLINICAL TRIAL: NCT01303887
Title: Purine-Alkylator Combination In Follicular Lymphoma Immuno-Chemotherapy for Older Patients: a Phase III Comparison of First-line R-CVP Versus R-FC
Brief Title: A Trial Looking at Rituximab and Chemotherapy as a Treatment for Follicular Lymphoma in Elderly Patients
Acronym: PACIFICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); Cancer Research UK (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ISRCTN99217456; 2008-004759-31 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Follicular Lymphoma
Keywords: PACIFICO; Follicular Lymphoma; Non-Hodgkin's Lymphoma; Rituximab; R-CVP; R-FC; Older
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Rituximab; Cyclophosphamide; Vincristine; Prednisolone; Methylprednisolone; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-CVP (Active Comparator): Repeated every 21 days for up to 8 cycles with response assessment after 4 cycles. Responders (PR/CR) after 8 cycles will receive Rituximab maintenance therapy for 2 years (12 bi-monthly cycles).
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisolone
- R-FC (Experimental): Repeated every 21 days for 4 cycles. Responders (PR/CR) after 4 cycles will receive 4 further cycles of Rituximab only. Responders after 8 cycles will receive Rituximab maintenance therapy for 2 years (12 bi-monthly cycles).
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m2 IV day 1,repeated every 21 days for 8 cycles. All patients who have achieved a CR or PR to induction therapy will receive rituximab maintenance (375mg/m2 every 2 months for 2 years).
  Other Names: Mabthera
  Arms: R-CVP
Drug: Cyclophosphamide — Cyclophosphamide 250mg/m2 PO day 1-3, repeated every 21 days for 4 (R-FC) or 8 cycles (R-CVP)
  Other Names: Cyclophosphamide monohydrate
Drug: Vincristine — Vincristine 1.4mg/m2 IV day 1,repeated every 21 days for 8 cycles.
  Other Names: vincristine sulfate
  Arms: R-CVP
Drug: Prednisolone — Prednisolone 40mg/m2 PO day 1-5, repeated every 21 days for 8 cycles.
  Other Names: Deltacortril
  Arms: R-CVP
Drug: Fludarabine — Fludarabine 40mg/m2 PO day 1-3,repeated every 21 days for 4 cycles
  Other Names: Fludara
  Arms: R-FC

SUMMARY:
The purpose of this study is to determine whether R-FC is more beneficial that R-CVP in the treatment of older patients (aged 60 or over) with Follicular Lymphoma (FL).

DETAILED DESCRIPTION:
FL predominantly affects the elderly, yet the optimum treatment for older patients with the disease has not been defined. The present study aims to address this question by comparing the drug combination that is currently considered the gold-standard (R-CVP) with a newer combination (R-FC) that might be more effective without being significantly more toxic. In order to take into account the balance between efficacy and toxicity, a dual primary endpoint has been employed: progression-free survival and toxicity in the form of grade 3-4 infection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma (grade 1,2, and 3a with material available for central review)
* Ann Arbor stage II-IV
* Aged 60 years or over, or aged less than 60 but anthracycline-based therapy contra-indicated
* No prior systemic therapy (one episode of prior local radiotherapy is allowed)
* At least one of the following criteria for initiation of treatment:
* Rapid generalized disease progression in the preceding 3 months
* Life threatening organ involvement
* Renal or macroscopic liver infiltration
* Bone lesions
* Presence of systemic symptoms or pruritus
* Haemoglobin < 10 g/dL or WBC < 3.0 × 109/L or platelet counts < 100 × 109/L due to marrow involvement
* Adequate haematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow):
* Haemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Written Informed Consent

Exclusion Criteria:

* Overt transformation to diffuse large B-cell lymphoma
* Grade 3b follicular lymphoma
* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningitis)
* WHO performance status 3 or 4
* Impaired renal function defined as estimated Glomerular filtration rate (eGFR) < 30 mL/min using the Modification of Diet in Renal Disease (MDRD) formula
* Impaired hepatic function defined as serum bilirubin more than twice upper limit of normal (unless due to lymphoma or Gilbert's syndrome)
* Life expectancy less than 12 months
* Pre-existing neuropathy
* Active auto-immune haemolytic anaemia
* Serological evidence of infection with HIV, hepatitis B (positivity for surface antigen or core antibody) or hepatitis C
* Allergy to murine proteins
* Corticosteroid treatment during the last 4 weeks, unless administered at a dose equivalent to no more than prednisolone 20mg/day continuously or a single course of prednisolone 1 mg/kg for up to 7 days
* Concomitant malignancies except adequately treated localised non-melanoma skin cancer or adequately treated in situ cervical cancer, or cancers that have been in remission for at least 5 years following surgery with curative intent.
* Major surgery (excluding lymph node biopsy) within 28 days prior to randomisation
* Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease)
* Treatment within a clinical trial within 30 days prior to trial entry
* Any other co-existing medical or psychological condition that will preclude participation in the study or compromise ability to give informed consent
* Adult patient under tutelage (not competent to sign informed consent)
* Pregnant or lactating women
* All men or women of reproductive potential, unless using at least two contraceptive precautions, one of which must be a condom

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Toxicity | 36 months
  The second primary outcome measure is grade 3-4 infection occurring anytime from the start of treatment until 6 months following the last dose of treatment, and this will be used as the toxicity end-point. Toxicity will be measured according to standard National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 following each cycle of treatment and at each subsequent follow-up visit until 6 months following the last dose of treatment.
Progression-free survival | 30 months

SECONDARY OUTCOMES:
Response rates (overall, complete and partial) following initial therapy | 24 weeks
Response rates following maintenance therapy | 30 months
Response duration | 30 months
Overall survival | End of study
Time to next treatment | End of study
Rate of large cell transformation | End of study
Response to second-line therapy | 30 months
Number of treatment cycles delivered | 30 months
Cumulative dose of individual drugs administered | 30 months
Quality of life | End of study
Cost effectiveness | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pettitt, Professor, Principal Investigator — University of Liverpool and Royal Liverpool and Broadgreen University Hospitals Trust
Locations (73):
- United Kingdom (73):
  - Aberdeen Royal Infirmary, Aberdeen
  - Ysbyty Gwynedd, Bangor
  - Birmingham Heartlands, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Frenchay Hospital, Bristol
  - Queen's Hospital, Burton, Burton-on-Trent
  - Addenbrookes Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - Velindre Hospital, Cardiff
  - Countess of Chester, Chester
  - Leighton Hospital, Crewe
  - Trafford General Hospital, Davyhulme
  - Russels Hall Hospital, Dudley
  - Royal Devon & Exeter Hospital, Exeter
  - Falkirk & District Royal Infirmary, Falkirk
  - Queen Elizabeth Hospital, Gateshead
  - Medway Maritime Hospital, Gillingham
  - Beatson Oncology Centre, Glasgow
  - Royal Alexandra Hospital, Glasgow
  - Harrogate District Foundation Trust, Harrogate
  - Northwick Park Hospital, Harrow
  - Princess Royal Hospital, Bromley, Hayes
  - Huddersfield Royal Infirmary, Huddersfield
  - Castle Hill Hospital, Hull
  - Raigmore Hospital,, Inverness
  - Ipswich Hospital, Ipswich
  - Kettering General Hospital, Kettering
  - The Queen Elizabeth Hospital, Kings Lynn, Kings Lynn
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - Guys & St Thomas Hospital, London
  - Kings College Hospital, London
  - Royal Free Hospital, London
  - St Bartholomews Hospital, London
  - University College Hospital, London
  - Altnagelvin Hospital, Londonderry
  - Luton & Dunstable Hospital, Luton
  - Kent Oncology Centre, Maidstone
  - Manchester Royal Infirmary, Manchester
  - The Christie Hospital, Manchester
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Northampton General Hospital, Northampton
  - Mount Vernon Hospital, Northwood
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Whiston Hospital, Prescot
  - Queens Hospital, Romford
  - Salford Royal Hospital, Salford
  - Salisbury District Hospital, Salisbury
  - Diana Princess of Wales Hospital, Scunthorpe
  - Royal Hallamshire Hospital, Sheffield
  - Wexham Park Hospital, Slough
  - South Tyneside District General Hospital, South Shields
  - Basingstoke and North Hampshire Hospital, Southampton
  - Southampton General Hospital, Southampton
  - St Richards Hospital, Southampton
  - Glan Clwyd Hospital, St Asaph
  - Stafford District General Hospital, Stafford
  - Lister Hospital, Stevenage
  - Sunderland Royal Hospital, Sunderland
  - Great Western Hospital, Swindon
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Hillingdon Hospital, Uxbridge
  - Pinderfields General Hospital, Wakefield
  - West Herts, Watford
  - Worcestershire Acute Hospitals NHS Trust, Worcester
  - Worthing Hospital, Worthing
  - York District Hospital, York

REFERENCES:
- See also: Cancer Research UK — http://www.cancerhelp.org.uk/trials/trials-search/trial-looking-rituximab-chemotherapy-treatment-follicular-lymphoma-elderly-patients-pacifico